CLINICAL TRIAL: NCT01870752
Title: Autologous Orthotopic Transplantation of Previously Cryopreserved Ovarian Tissue
Brief Title: Ovarian Tissue Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02813
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Infertile Females or Females With Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: Thaw and surgical transplantation of previously collected cryopreserved ovarian cortical tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transplantation of previously cryopreserved ovarian tissue (Other): Surgical transplantation of previously collected cryopreserved ovarian cortical tissue.
  Interventions: Procedure: Transplantation of previously cryopreserved ovarian tissu

INTERVENTIONS:
Procedure: Transplantation of previously cryopreserved ovarian tissu

SUMMARY:
Chemotherapy and radiation therapy for the treatment of cancer can compromise fertility. Ovarian tissue cryopreservation is an experimental strategy offered at The University of Pennsylvania to preserve future fertility (protocol 806062). The primary objective of this study is to determine the efficacy and safety of autologous transplantation of previously cryopreserved ovarian cortical tissue in patients who experience infertility or ovarian insufficiency after cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* Female patient between the ages of 18 and 45 years
* Previously cryopreserved and stored cortical ovarian tissue available for autologous transplantation
* Ovarian insufficiency defined as an elevated FSH over 10
* Inability to conceive after 6 months of unprotected intercourse with male
* Reasonably good health
* Candidate for pregnancy
* Written clearance for the procedure from the patients oncologist

Exclusion Criteria:

* Patients considered to be high risk for surgical complications will be excluded from the research protocol
* Women who are known to be positive for the BRCA mutation
* Women with a history of leukemia, ovarian cancer or a cancer that likely involved the ovaries at the time of ovarian tissue collection
* Women with psychological, psychiatric, or other conditions which prevent giving fully informed consent
* Current pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy | 5 years
Return of menstrual function | 5 years

SECONDARY OUTCOMES:
Cancer recurrence | 5 years
Surgical Complications of ovarian tissue transplantation | 5 years
  Including infection, hospital readmission, re-operation
Acceptability | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa R Gracia, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States